CLINICAL TRIAL: NCT02996877
Title: Outcomes of Percutaneous Revascularization for Management of Surgically Ineligible Patients With Multivessel or Left Main Coronary Artery Disease: A Prospective Registry
Brief Title: Outcomes of Surgically Ineligible Patients With Multivessel CAD
Acronym: OPTIMUM
Status: Completed | Type: Observational
Sponsor: Saint Luke's Health System (Other)
Collaborators: Piedmont Heart Institute, Inc., Atlanta, GA (Industry)
Responsible Party: Sponsor
Other Study IDs: ISROTH10299
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Guideline Directed Medical Therapy: Patients who have an initial treatment strategy of using guideline-directed medical therapy only.
- Percutaneous Coronary Intervention: Patients who will have a Percutaneous Coronary Intervention as the initial treatment strategy along with guideline directed medical therapy.

SUMMARY:
The OPTIMUM registry is a minimal risk observational study that uses a prospective cohort design to follow patients who have multivessel or left main coronary artery disease ("surgical anatomy" according to ACC/AHA Appropriateness Criteria for PCI12) and are deemed ineligible for coronary artery bypass surgery. It is anticipated that 20 sites will be selected to participate in the registry from a national network of leading centers across the United States with recognized expertise in both complex PCI and coronary artery bypass surgery. We will invite leading cardiac centers, as defined by US News and World reports rankings for heart care. Additional sites may be added to meet the target enrollment goal.

DETAILED DESCRIPTION:
Objectives 1. Compare 30-day mortality and the composite of mortality and morbidity following high-risk percutaneous coronary revascularization with predicted Society of Thoracic Surgeons (STS) survival and morbidity in patients with severe multivessel or left main coronary artery disease (CAD).

2. Compare the 12-month health status and clinical outcomes of surgically ineligible multivessel or left main CAD patients treated with PCI compared to those treated with a medical therapy alone.

3. Understand the association between completeness of revascularization and long-term health status and clinical outcomes among patients with multivessel or left main CAD treated with PCI deemed ineligible for surgery.

4. Compare 6-month and 1-year survival among surgically ineligible high-risk PCI patients with predicted STS survival (ASCERT risk model)

5. Determine the justification for surgical ineligibility by cardiologists and cardiac surgeons among patients with severe multivessel or left main coronary artery disease (CAD).

6. Describe the frequency and predictors of PCI versus medical management among surgically ineligible patients with severe multivessel or left main CAD.

7. Describe the frequency and predictors of complete revascularization in this population.

8. Describe the costs and costs per quality adjusted life year (QALY) gained of the strategy of management of multivessel or left main CAD with PCI versus medical therapy among surgically ineligible patients.

ELIGIBILITY:
Inclusion Criteria:

- Participant Selection Inclusion Criteria

1. Participant undergoes coronary angiography revealing unprotected left main stenosis of > 50%, 3 vessel disease with stenoses > 70% or 2 vessel coronary disease (>70%) with one lesion involving the proximal LAD. Patients will also be included if there is FFR evidence of flow limiting stenosis (FFR ≤ 0.80) in the setting of > 40% angiographic stenosis the left main, 3 epicardial coronaries or 2 vessels including the proximal LAD. Patients with prior bypass surgery will be included if they have ≥ 2 epicardial vascular distributions subtended by a severe native coronary stenosis with either no bypass graft supplying the vessel, a severely diseased (>70% stenosis) bypass graft supplying the affected vessel or an occluded bypass graft to the affected vessel.
2. Patient considered high risk for coronary artery bypass surgery and declared ineligible for surgery by the heart team.
3. Patient is experiencing clinical symptoms consistent with obstructive coronary artery disease or with evidence of coronary ischemia on non-invasive/invasive (FFR) functional testing.
4. Subject is ≥ 18 years of age at the time of consent and is willing to sign an informed consent document approved by the enrolling hospital's Institutional Review Board and follow-up for 12-months following enrollment in the study
5. Patient is able to speak English.

Exclusion Criteria:

* Exclusion Criteria

  1. Established iodine allergy that cannot be managed medically, allergy to everolimus, or absolute contraindication to aspirin, P2Y12 antagonist therapy with either clopidogrel, prasgurel, ticagrelor or ticlopidine or absolute contraindication to bivalirudin and heparin precluding procedural anticoagulation.
  2. Emergent revascularization required for ST-elevation myocardial infarction or cardiac arrest, or severe sustained hemodynamic instability.
  3. Patients presenting late after STEMI (> 12 hours after symptom onset) for "salvage" PCI.
  4. Too hard of hearing to do follow-up by telephone.
  5. Currently incarcerated.
  6. Dementia.
  7. Subjects with no way to be contacted by telephone for follow-up, including those who live outside of the U.S. or spend significant time outside of the U.S.
  8. Patients with conditions such as cancer, mental illness, or other pathology which, in the opinion of the local investigator, might put the patient at risk, preclude follow-up or confound the results of the study.
  9. Patients who refuse.
  10. Female subjects with a positive quantitative or qualitative pregnancy test will not be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients identified as having Coronary Artery Disease with Left Main or multivessel involvement, who have been deemed ineligible to receive coronary bypass surgery as treatment.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
30 day survival following high risk percutaneous coronary revascularization who are at high risk. | 30 days
  Patients will be followed with phone calls at 30 days.

SECONDARY OUTCOMES:
12 month Seattle Angina Questionnaire Overall summary score comparing patients undergoing PCI versus those treated with medical therapy only. | 12 months
  Patients will be called at 12 months time by the centralized follow up center.

CONTACTS AND LOCATIONS:
Overall Officials: Adam C Salisbury, MD MSc, Principal Investigator — Saint Luke's Health System; David E Kandzari, MD, Principal Investigator — Piedmont Heart and Vascular Institute; James A Grantham, MD, Principal Investigator — Saint Luke's Health System
Locations (21):
- United States (21):
  - Banner University Medical Center, Phoenix, Arizona
  - Unifersity of California San Diego Medical Center, San Diego, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University in Saint Louis, St Louis, Missouri
  - Northwell Health System, Manhasset, New York
  - Columiba University Medical Center, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Geisinger Health System, Danville, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Virginia Medical Center, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Charleston Area Medical Center, Charleston, West Virginia